CLINICAL TRIAL: NCT03294499
Title: Positive Attitudes Concerning Infant Feeding- a Questionnaire for Women Living With HIV
Acronym: PACIFY
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 17IC3795; 221592 (Other: IRAS)
Record Dates: First submitted 2017-08-01; First posted 2017-09-27 (Actual); Results first posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2022-05

CONDITIONS: Human Immunodeficiency Virus
Keywords: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Patients will be asked to complete one off questionnaire.

SUMMARY:
The PACIFY Study is a questionnaire for antenatal(third trimester) and postnatal(three months post delivery) Human Immunodeficiency Virus (HIV) positive women attending clinics in London and Brighton. The current World Health Organisation guidance advises HIV positive women, who are adhering to antiretroviral therapy (ART), to exclusively breastfeed for the first 6 months of the infant's life and continue supplemental breastfeeding for up to 2 years.

This is conflicts with the current British HIV Association guidelines which advise exclusive formula feeding. The reason for this difference is the relative safety of formula feeding in the United Kingdom(UK)against the low but persisting risk of HIV infection through breast-feeding. The aim of the PACIFY study is to explore attitudes towards breastfeeding amongst HIV positive women, who are either pregnant or post-partum. The study will also assess the understanding of current infant feeding guidance by these women and assess their current or recent infant feeding practice. It will also look at whether HIV positive mothers would be willing and able to comply with special monitoring and guidance whilst breastfeeding if the guidelines were to change. The study aims to analyse 100 questionnaires completed over a 3-6 month period.

DETAILED DESCRIPTION:
All eligible female patients (currently or recently pregnant) attending routine HIV-related appointments will be invited to participate and a participant information sheet will be given. Those who have consented to join the study will be given a short questionnaire to complete and return during that attendance. The questionnaire takes about 15 minutes to complete. The option of returning the questionnaire by post will be available but not encouraged.

During the collection period, women with HIV attending either antenatal (third trimester) or postnatal (within three months of delivery) care will be eligible to participate, but they will only be asked once, either before or after delivery.

Ideally equivalent numbers of pre and postnatal participants will be enrolled. Participants given a questionnaire and have a centre and unique study number. Maternal cluster of differentiation 4 (CD4) count and HIV Viral load nearest to time of questionnaire completion will be recorded if patient consents.

Participants will be able to place their completed paper questionnaires in a sealed envelope in a box in the clinic.Participants will be informed that their questionnaire responses will not be seen by clinical staff (unless participants request staff support in completion of the questionnaire) or recorded in their clinical notes. In the clinics the study log will be the only document linking study number with hospital identification (ID)number and soundex. Completed questionnaires will be stored securely in local sites prior to transfer to St Mary's Hospital (by the study team). The study log will be maintained securely along with the delegation log by the site lead investigator.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Able to give written informed consent
* Post-natal and antenatal HIV positive women

Exclusion Criteria:

* Age <18 years
* Patients who are unable to consent.
* Women with HIV who have not been pregnant.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This is a questionnaire for HIV positive women who are in their third trimester and three months post partum
Study Population: HIV positive women who are three months post partum and third trimester
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hermione Lyall, MBChB, Study Chair — Imperial College Healthcare NHS Trust
Locations (10):
- United Kingdom (10):
  - Brighton and Sussex NHS Trist, Brighton
  - Barts Health NHS Trust, London
  - CENTRAL AND NORTH WEST London NHS Trsut, London
  - Chelsea and Westminister NHS Trust, London
  - Guys and St Thomas NHS Trust, London
  - Homerton University Hospital Nhs Trust, London
  - Imperial College Healthcare NHS Trust, London
  - Kings College NHS Trust, London
  - Lewisham and Greenwich NHS Trust, London
  - London Northwest Healthcare NHS Trust, London

IPD SHARING:
Plan to Share IPD: No
Results will be presented at a conference and published.

REFERENCES:
- [Result] Nyatsanza F, Gubbin J, Gubbin T, Seery P, Farrugia P, Croucher A, Gilleece Y, Rosenvinge M, Roedling S, Sarner L, Nayagam D, Stradling C, Namiba A, Fearnley N, Lyall H. Over a third of childbearing women with HIV would like to breastfeed: A UK survey of women living with HIV. Int J STD AIDS. 2021 Aug;32(9):856-860. doi: 10.1177/0956462421999951. Epub 2021 Feb 25. PMID 33629917

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient were recruited from medical outpatient clinics across England The study period was May 2017 -May 2018
Groups:
- Women Living With HIV: Women were in their third trimester or three months post-partum
Period: Overall Study
Arm/Group | Women Living With HIV
Started | 94
Completed | 94
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 94 participants were recruited from 12 clinics in England
Groups:
- Women Living With HIV: The PACIFY was a descriptive questionnaire with no study arms Patients were recruited from 12 clinics in England.Participant were asked to complete a six paged questionnaire which would be analysed.
Arm/Group | Women Living With HIV
Number analyzed (Participants) | 94
Age, Categorical [Count of Participants; unit: Participants] — Descriptive Questionnaire
  Participants
    <=18 years | 0
    Between 18 and 65 years | 94
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 72
  White | 10
  More than one race | 3
  Unknown or Not Reported | 0
Immigration [Count of Participants; unit: Participants]
  Immigrants | 70
  Non-immigrants | 18
  No answer | 6
Employment status [Count of Participants; unit: Participants]
  Employed | 51
  Unemployed | 43
Education status [Count of Participants; unit: Participants]
  Higher education | 77
  Secondary school | 13
  Primary school | 3
  No answer | 1
HIV diagnosed [Count of Participants; unit: Participants]
  Before pregnancy | 71
  During current pregnancy | 23
HIV parameters [Count of Participants; unit: Participants]
  HIV viral load <50 copies/ml | 86
  HIV viral load >50 copies/ml | 1
  No answer | 7

OUTCOME MEASURES:

1. Primary Outcome: Knowledge and Experiences of Breastfeeding Among Women Living With HIV
Description: Participants were recruited by clinicians from 12 HIV clinics across England (South East, West Midlands and West Yorkshire) between June 2017 and June 2018. Participants were given the study patient information leaflet and consent form when they attended their regular pre- or postnatal outpatient appointment and, if they agreed to participate, they completed the anonymised questionnaire (Supplemental Appendix X) during the same visit. All the questionnaires were collated at Imperial College Healthcare NHS Trust.
  In the data table, breastfeeding has been abbreviated to BF.
Time Frame: At their pre-or postnatal outpatient appointment, an average of one day
Measure: Count of Participants; unit: Participants
Arm/Group | Women Living With HIV
Number analyzed (Participants) | 94
Participants
  Have any friends, family or community members questioned you about your reasons for not BF?: Yes | 58
  Have any friends, family or community members questioned you about your reasons for not BF?: No | 25
  Have any friends, family or community members questioned you about your reasons for not BF?: Don't know | 0
  Have any friends, family or community members questioned you about your reasons for not BF?: No answer | 11
  Have you ever had to lie about your reasons for not BF?: Yes | 62
  Have you ever had to lie about your reasons for not BF?: No | 21
  Have you ever had to lie about your reasons for not BF?: Don't know | 0
  Have you ever had to lie about your reasons for not BF?: No answer | 11
  If you did not have HIV, would you BF your child?: Yes | 84
  If you did not have HIV, would you BF your child?: No | 2
  If you did not have HIV, would you BF your child?: Don't know | 8
  If you did not have HIV, would you BF your child?: No answer | 0
  Living with HIV, would you like to BF your child?: Yes | 36
  Living with HIV, would you like to BF your child?: No | 45
  Living with HIV, would you like to BF your child?: Don't know | 6
  Living with HIV, would you like to BF your child?: No answer | 7
  Do you think it's safe for women with detectable HIV in the blood to BF?: Yes | 3
  Do you think it's safe for women with detectable HIV in the blood to BF?: No | 63
  Do you think it's safe for women with detectable HIV in the blood to BF?: Don't know | 22
  Do you think it's safe for women with detectable HIV in the blood to BF?: No answer | 6
  Do you think it's safe for women on treatment with fully suppressed HIV to BF?: Yes | 26
  Do you think it's safe for women on treatment with fully suppressed HIV to BF?: No | 33
  Do you think it's safe for women on treatment with fully suppressed HIV to BF?: Don't know | 31
  Do you think it's safe for women on treatment with fully suppressed HIV to BF?: No answer | 4
  If you were to BF, would you have monthly blood tests to check your viral load stays undetectable?: Yes | 83
  If you were to BF, would you have monthly blood tests to check your viral load stays undetectable?: No | 10
  If you were to BF, would you have monthly blood tests to check your viral load stays undetectable?: Don't know | 0
  If you were to BF, would you have monthly blood tests to check your viral load stays undetectable?: No answer | 1
  If you were to BF, would you be willing for your baby to have a monthly HIV blood test?: Yes | 79
  If you were to BF, would you be willing for your baby to have a monthly HIV blood test?: No | 13
  If you were to BF, would you be willing for your baby to have a monthly HIV blood test?: Don't know | 0
  If you were to BF, would you be willing for your baby to have a monthly HIV blood test?: No answer | 2
  Do you have any concerns about BF while you are taking anti-HIV medicines?: Yes | 47
  Do you have any concerns about BF while you are taking anti-HIV medicines?: No | 44
  Do you have any concerns about BF while you are taking anti-HIV medicines?: Don't know | 1
  Do you have any concerns about BF while you are taking anti-HIV medicines?: No answer | 2
  Have you heard of 'exclusive BF' (giving the baby breast milk only and no other feeds or drinks)?: Yes | 63
  Have you heard of 'exclusive BF' (giving the baby breast milk only and no other feeds or drinks)?: No | 29
  Have you heard of 'exclusive BF' (giving the baby breast milk only and no other feeds or drinks)?: Don't know | 0
  Have you heard of 'exclusive BF' (giving the baby breast milk only and no other feeds or drinks)?: No answer | 2
  If you were to BF, would you be happy to exclusively BF?: Yes | 51
  If you were to BF, would you be happy to exclusively BF?: No | 41
  If you were to BF, would you be happy to exclusively BF?: Don't know | 0
  If you were to BF, would you be happy to exclusively BF?: No answer | 2
  Have any healthcare workers discussed BF with you?: Yes | 84
  Have any healthcare workers discussed BF with you?: No | 8
  Have any healthcare workers discussed BF with you?: Don't know | 0
  Have any healthcare workers discussed BF with you?: No answer | 2
  Would you like more information on the benefits and disadvantages of BF?: Yes | 45
  Would you like more information on the benefits and disadvantages of BF?: No | 48
  Would you like more information on the benefits and disadvantages of BF?: Don't know | 0
  Would you like more information on the benefits and disadvantages of BF?: No answer | 1

2. Primary Outcome: Views on Infant Feeding for Women Living With HIV
Description: The PACIFY study (Positive Attitudes Concerning Infant Feeding) sought to explore the views, concerns and issues surrounding breastfeeding in women living with HIV (WLHs).
  Questions within the questionnaire:
  1. If you did not have HIV, would you breastfeed your child?
  2. Living with HIV, would you like to breastfeed your child?
Time Frame: At their pre-or postnatal outpatient appointment, an average of one day
Measure: Number; unit: percentage of total participants
Groups:
- Women Living With HIV: The PACIFY was a descriptive questionnaire with no study arms
Arm/Group | Women Living With HIV
Number analyzed (Participants) | 94
percentage of total participants
  would like to breastfeed if they were HIV negative | 89
  would like to breastfeed while living with HIV | 38

ADVERSE EVENTS:
Time Frame: Data was collected over a 12 month period
Groups:
- PACIFY Study: They were no adverse events reported
Arm/Group | PACIFY Study
All-Cause Mortality (participants affected / at risk) | 0/94
Serious Adverse Events (participants affected / at risk) | 0/94
Other Adverse Events (participants affected / at risk) | 0/94

LIMITATIONS AND CAVEATS:
We sampled a small number of participants and we were unable to ascertain how many participants refused to respond to questionnaire

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-01-23): https://cdn.clinicaltrials.gov/large-docs/99/NCT03294499/Prot_SAP_ICF_000.pdf